CLINICAL TRIAL: NCT04288999
Title: JCOG1801: A Phase III Randomized Controlled Trial Comparing Surgery Plus Adjuvant Chemotherapy With Preoperative Chemoradiotherapy Followed by Surgery Plus Adjuvant Chemotherapy for Locally Recurrent Rectal Cancer (RC-SURVIVE Study)
Brief Title: Surgery Plus Chemo Versus Chemoradiotherapy Followed by Surgery Plus Chemo for Locally Recurrent Rectal Cancer
Acronym: JCOG1801
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Center Hospital East (Other)
Collaborators: Japan Clinical Oncology Group (Other); Japan Agency for Medical Research and Development (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG1801
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Rectal Cancer Recurrent
Keywords: Rectal cancer; Locally recurrent rectal cancer; Chemoradiotherapy; Surgery; Chemotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Drug Therapy; Capecitabine; Radiotherapy; Methods; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Preoperative chemoradiotherapy (CRT) followed by Surgery plus Adjuvant chemotherapy
  Preoperative CRT: capecitabine (1650 mg/m2/day) and radiotherapy (50.4 Gy/28 Fr)
  Adjuvant chemotherapy: CAPOX (capecitabine+oxaliplatin) or mFOLFOX6 (5-fluorouracil+l-leucovorin+oxaliplatin) or capecitabine or 5-fluorouracil (FU) +l-leucovorin (LV)
  CAPOX: oxaliplatin (130 mg/m2/day, day 1) and oral capecitabine (2000 mg/m2/day, twice daily, days 1-14)
  mFOLFOX6: oxaliplatin 85 mg/m2 with l-LV 200 mg/m2 for over 2 hours followed by a fluorouracil 400 mg/m2 bolus and 2400 mg/m2 continuous infusion over 46 hours.
  Capecitabine: 2000 mg/m2/day, twice daily, days 1-14
  5-FU+l-LV: leucovorin 200 mg/m2 for over 2 hours followed by a fluorouracil 400 mg/m2 bolus and 2400 mg/m2 continuous infusion for over 46 hours
  Interventions: Drug: Chemotherapy; Radiation: Preoperative radiotherapy; Other: Procedure
- Arm B (Active Comparator): Surgery plus Adjuvant chemotherapy
  Adjuvant chemotherapy: CAPOX or mFOLFOX6 or capecitabine or 5-FU+l-LV
  CAPOX: oxaliplatin (130 mg/m2/day, day 1) and oral capecitabine (2000 mg/m2/day, twice daily, days 1-14)
  mFOLFOX6: oxaliplatin 85 mg/m2 with l-LV 200 mg/m2 for over 2 hours followed by a fluorouracil 400 mg/m2 bolus and 2400 mg/m2 continuous infusion over 46 hours.
  Capecitabine: 2000 mg/m2/day, twice daily, days 1-14
  5-FU+l-LV: leucovorin 200 mg/m2 for over 2 hours followed by a fluorouracil 400 mg/m2 bolus and 2400 mg/m2 continuous infusion for over 46 hours
  Interventions: Drug: Chemotherapy; Other: Procedure

INTERVENTIONS:
Drug: Chemotherapy — Adjuvant chemotherapy: CAPOX or mFOLFOX6 or capecitabine or 5-FU+l-LV
  CAPOX: oxaliplatin (130 mg/m2/day, day 1) and oral capecitabine (2000 mg/m2/day, twice daily, days 1-14)
  mFOLOX6: oxaliplatin 85 mg/m2 with l-LV 200 mg/m2 for over 2 hours followed by a fluorouracil 400 mg/m2 bolus and 2400 mg/m2 continuous infusion over 46 hours.
  Capecitabine: 2000 mg/m2/day, twice daily, days 1-14
  5-FU+l-LV: leucovorin 200 mg/m2 for over 2 hours followed by a fluorouracil 400 mg/m2 bolus and 2400 mg/m2 continuous infusion for over 46 hours
  Other Names: CAPOX or mFOLFOX6 or capecitabine or 5-FU+l-LV
Radiation: Preoperative radiotherapy — Preoperative chemoradiotherapy (CRT) followed by Surgery plus Adjuvant chemotherapy
  Preoperative CRT: capecitabine (1650 mg/m2/day) and radiotherapy (50.4 Gy/28 Fr)
  Other Names: Capecitabine plus radiotherapy
  Arms: Arm A
Other: Procedure — Surgery for Locally Recurrent Rectal Cancer (LRRC) will be performed within 42 days from registration for the patients in arm A, and between days 56 and 98 from the completion of the preCRT for the patients in arm B.
  Appropriate surgical procedure will be performed to achieve R0 resection, such as low anterior resection, super low anterior resection, intersphincteric resection, Hartmann procedure, rectal amputation, pelvic exenteration, tumor resection, or lateral lymph node dissection
  Other Names: Surgery

SUMMARY:
JCOG1801 is a randomized phase III trial which was initiated in Japan in August 2019 to confirm the superiority of preoperative chemoradiotherapy followed by surgery plus adjuvant chemotherapy for local relapse-free survival over standard treatment, i.e. surgery plus adjuvant chemotherapy, for previously non-irradiated locally recurrent rectal cancer.

DETAILED DESCRIPTION:
In all, 110 patients from 43 Japanese institutions will be recruited over a period of 6 years. Eligible patients would be registered and randomly assigned to each group with an allocation ratio of 1:1. The primary endpoint is local relapse-free survival. The secondary endpoints are overall survival, relapse-free survival, proportion of local relapse, proportion of distant relapse, proportion of patients with pathological R0 resection, response rate of preoperative chemoradiotherapy (preoperative chemoradiotherapy arm), pathological complete response rate (preoperative chemoradiotherapy arm), proportion of patients who completed the protocol treatment, incidence of adverse events (adverse reactions), and quality of life after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically proven adenocarcinoma or adenosquamous carcinoma on the resected specimen of the initial rectal cancer or endoscopic biopsy from the initial rectal cancer.
2. The main tumor location of the initial rectal cancer is upper, middle or lower rectum, or anal canal.
3. Either of the following treatments was performed for the initial rectal cancer, and classified as R0/1 or ER (Endoscopical R)0/1 on pathological diagnosis.

   i) Surgical resection (including local resection, with or without lymph node dissection).

   ii) Endoscopic resection.
4. Patients with distant metastasis during or after treatment for the initial rectal cancer, and radical surgical resection or radical radiotherapy performed more than 168 days before registration is eligible.
5. Recurrent rectal cancer diagnosed by any of the following modalities after treatment for the initial rectal cancer.

   i) The recurrent lesion is pathologically diagnosed. ii) Diagnosed as local recurrence by more than two modalities among contrast-enhanced CT, contrast-enhanced MRI, or positron emission computed tomography (PET).

   iii) Chronological progression of the lesion seen on more than one modality among contrast-enhanced CT, MRI, or PET.
6. The main tumor location is within pelvis as seen on contrast-enhanced CT and MRI if recurrent lesion is multiple, or recurrent lesions spread outside of pelvis continuously.
7. LRRC is diagnosed with no following condition. i) Judged as resectable endoscopically. ii) Depth of invasion within the muscularis propria as seen on contrast-enhanced CT, MRI, or PET in case of recurrence inside the intestine iii) Solitary ovarian metastasis. iv) Recurrence of the common iliac lymph node alone.
8. LRRC is diagnosed as resectable, and all the following conditions must be fulfilled:

   i) No distant metastasis on contrast-enhanced CT (cM0). ii) Estimated circumferential resection margin >0 mm. iii) Leg amputation not required. iv) Preservation of the first sacral nerve possible.
9. No prior surgery for recurrent rectal cancer.
10. No prior pelvic irradiation for any malignancies.
11. A patient who has received systemic chemotherapy for any malignancies and the final dose was administered more than 14 days ago.
12. Age at registration is 20 to 80 years old.
13. Eastern Cooperative Oncology Group (ECOG) performance status is 0 or 1.
14. Measurable lesion is not mandatory.
15. Adequate oral intake.
16. Sufficient organ function. i) Neutrophil count >= 1,500/mm3 ii) Hemoglobin >= 9.0 g/dL iii) Platelet count >= 100,000/mm3 iv) Total Bilirubin =< 2.0 mg/dL v) Aspartate aminotransferase (AST) =< 100 U/L vi) Alanine Aminotransferase (ALT) =< 100 U/L vii) Cr =< 1.5 mg/dL
17. Open surgery or laparoscopic surgery is planned.
18. Written informed consent is obtained.

Exclusion Criteria:

1. Synchronous or metachronous (within 5 years) malignancies except cancer with 5-year relative survival rate of 95% or more such as carcinoma in situ, intramucosal tumor, or early stage cancers.
2. Infections requiring systemic treatment.
3. Body temperature higher than 38 degrees Celsius at registration.
4. Pregnant female, female within 28 days post-parturition, or lactating mother. Men with partners planning conception in the near future.
5. Severe psychological disease.
6. Continuous systemic corticosteroid or immunosuppressant treatment.
7. Uncontrollable diabetes mellitus.
8. Uncontrollable hypertension.
9. Unstable angina pectoris, or history of myocardial infarction within 6 months.
10. Uncontrollable valvular disease, dilated cardiomyopathy, or hypertrophic cardiomyopathy.
11. Positive serum Hepatitis B (HB)s antigen or serum Hepatitis C Virus (HCV) antibody.
12. Positive serum HIV antibody.
13. Interstitial pneumonia, pulmonary fibrosis, or severe emphysema on chest CT.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Locally recurrent free survival | 3-years after registration
  the period from registration in the trial to either the first event of local relapse or death from any cause and censored at the last date of contact for a living patient

SECONDARY OUTCOMES:
Overall survival (OS) | 3-years after registration
  s the time from registration to death from any cause and censored at the last date of contact for a living patient
Recurrence free survival (RFS) | 3-years after registration
  the time from registration to either the first incidence of relapse or death from any cause and censored at the last date of contact for a living patient
Local relapse rate | 3-years after registration
  Proportion of local relapse
Distant relapse rate | 3-years after registration
  Proportion of distant relapse
R0 resection rate | 1 month after surgery
  Proportion of patients with pathological R0 resection
Response rate of preoperative chemoradiotherapy (preCRT) | before surgery
  Response rate of preCRT (arm B)
Pathological complete response rate | 1 month after surgery
  Pathological complete response rate (arm B)
Completeness of the protocol treatment | 8 months after surgery
  Proportion of patients who completed the protocol treatment
Adverse event rate | 3-years after surgery registration
  Incidence of adverse events (adverse reactions)
QOL | 3-years after registration
  QOL after surgery based on the Trial Outcome Index-Physical/Functional/Colorectal (TOI-PFC) [0(better)-84(worse)]

CONTACTS AND LOCATIONS:
Overall Officials: Masaaki Ito, MD, PhD, Principal Investigator — National Cancer Center Hospital East
Locations (45):
- Japan (45):
  - Chiba Cancer Center, Chiba
  - Gifu University School of Medicine, Gifu
  - Saitama Medical University International Medical Center, Hidaka
  - Kansai Medical University Hospital, Hirakata
  - Hiroshima City Asa Citizens Hospital, Hiroshima
  - Hiroshima City Hospital, Hiroshima
  - Shimane University Faculty of Medicine, Izumo
  - Ishikawa Prefectural Central Hospital, Kanazawa
  - National Cancer Center Hospital East, Kashiwa
  - Saitama Medical Center, Saitama Medical University, Kawagoe
  - Kochi Health Sciences Center, Kochi
  - Kumamoto University Hospital, Kumamoto
  - Kurashiki Central Hospital, Kurashiki
  - Kurume University School of Medicine, Kurume
  - National Hospital Organization Shikoku Cancer Center, Matsuyama
  - Kyorin University Faculty of Medicine, Mitaka
  - Iwate Medical University, Morioka
  - Nagoya University Graduate School of Medicine, Nagoya
  - Niigata Cancer Center Hospital, Niigata
  - Hyogo College of Medicine, Nishinomiya
  - Okayama Saiseikai General Hospital, Okayama
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka City General Hospital, Osaka
  - Ogaki Municipal Hospital, Ōgaki
  - Gunma Prefectural Cancer Center, Ōta-ku
  - Saitama Cancer Center, Saitama
  - Sapporo-Kosei General Hospital, Sapporo
  - Miyagi Cancer Center, Sendai
  - Shizuoka Cancer Center, Shizuoka
  - Osaka University Graduate School of Medicine, Suita
  - Suita Municipal Hospital, Suita
  - Osaka Medical College, Takatsuki
  - National Defense Medical College, Tokorozawa
  - National Cancer Center Hospital, Tokyo
  - Toho University Ohashi Medical Center, Tokyo
  - Toho University Omori Medical Center, Tokyo
  - Tokyo Medical and Dental University Hospital, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - Tokyo Metropolitan Cancer and Infectious diseases Center Komagome Hospital, Tokyo
  - Tochigi Cancer Center, Utsunomiya
  - Yamagata Prefectural Central Hospital, Yamagata
  - Kanagawa Cancer Center, Yokohama
  - Saiseikai Yokohama-shi Nanbu Hospital, Yokohama
  - Yokohama City University Medical Center, Yokohama
  - Oita University Faculty of Medicine, Yufu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hashimoto T, Tsukada Y, Ito M, Kanato K, Mizusawa J, Fukuda H, Tsukamoto S, Takashima A, Kanemitsu Y. Utility of circulating tumour DNA for prognosis and prediction of therapeutic effect in locally recurrent rectal cancer: study protocol for a multi-institutional, prospective observational study (JCOG1801A1, CAP-LR study). BMJ Open. 2023 Aug 16;13(8):e073217. doi: 10.1136/bmjopen-2023-073217. PMID 37586869
- [Derived] Kadota T, Tsukada Y, Ito M, Katayama H, Mizusawa J, Nakamura N, Ito Y, Bando H, Ando M, Onaya H, Fukuda H, Kanemitsu Y. A phase III randomized controlled trial comparing surgery plus adjuvant chemotherapy with preoperative chemoradiotherapy followed by surgery plus adjuvant chemotherapy for locally recurrent rectal cancer: Japan Clinical Oncology Group study JCOG1801 (RC-SURVIVE study). Jpn J Clin Oncol. 2020 Aug 4;50(8):953-957. doi: 10.1093/jjco/hyaa058. PMID 32409830
- See also: Japan Registry of Clinical Trials — https://jrct.niph.go.jp/en-latest-detail/jRCTs031190076